CLINICAL TRIAL: NCT05305638
Title: Investigation of the Effect of Telerehabilitation-Based Physiotherapy Training on Respiration, Quality of Life, Physical Activity and Fatigue in Individuals With Covid-19
Brief Title: Tele-Rehabilitation in Individuals With Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Emine Nur Demircan, Specialist Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Covid-19
Record Dates: First submitted 2022-03-30; First posted 2022-03-31 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: Covid-19; Breathing; Quality of Life; Physical Activity; Fatigue
MeSH Terms: conditions — COVID-19; Respiratory Aspiration; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Exercise
- Control Group (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Home-based physical activity programs are very important to strengthen the immune system, which is extremely important in the fight against COVID-19 infection, and to protect physical and mental health. In addition, since the pulmonary rehabilitation sessions carry a high risk of transmission, it is recommended that the program be carried out with applications such as single-session training, tele-rehabilitation or home program. Although the home pulmonary rehabilitation program is adapted to the individual, it generally includes positioning, mobilization, relaxation exercises, respiratory training, respiratory muscle exercises, upper and lower extremity exercises, walking, climbing stairs and cycling exercises. The general opinion is that telerehabilitation practices have many benefits such as increasing the quality of life and physical activity. In addition to these benefits, telerehabilitation applications come to the fore in the Covid-19 period with its complementary feature.

SUMMARY:
Coronavirus Disease (COVID-19) is a respiratory disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-cov-2). This study was planned as a single-blind randomized controlled pilot study to compare the effectiveness of telerehabilitation-based exercise training applied to individuals with Covid-19. Individuals will be divided into two groups, the control group and the study group. All assessments will be made online twice, before and after treatment. Socio-demographic data of individuals who agreed to participate in the study, disease information about Covid-19, MRC Dyspnea Scale, COVID-19 Fear Scale, International Physical Activity Questionnaire-Short Form, ST. George Respiratory Questionnaire, Fatigue Severity Scale, Nottingham Health Profile will be questioned and recorded. The obtained data will be analyzed with statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* A score in the range of 0-3 on the MRC Dyspnea Scale.
* Not have any vestibular, orthopedic or neurological disease that will affect muscle strength, balance and coordination.
* Not having undergone surgery in the last 6 months.
* Not having undergone any surgical procedure that may affect the musculoskeletal system of the spinal column, lower extremities or upper extremities.
* It was being cooperative and volunteering.

Exclusion Criteria:

* Severe liver and kidney disease or new and progressive damage to liver and kidney function, deep vein thrombosis and pulmonary embolism, suspected aortic stenosis, having a disease/condition for which exercise is contraindicated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The Fear of COVID-19 Scale | baseline to 6 week after
  The Fear of COVID-19 Scale was used to measure the level of fear caused by Covid-19. Each question of the scale, which consists of 7 questions, is graded on a 5-point Likert scale (1- I strongly disagree. 5- I strongly agree). A high score indicates greater fear of Covid-19.
MRC Dyspnea Scale | baseline
  The MRC Dyspnea Scale was used to assess the participants' dyspnea levels. It is a five-point scale based on various physical exercises that produce a feeling of dyspnea. It consists of five items. The person's respiratory distress is graded from 0 (no shortness of breath) to 4 (shortness of breath during activities such as being confined to home and dressing).
International Physical Activity Questionnaire-Short Form | baseline to 6 week after
  The physical activity levels of the participants were evaluated with the International Physical Activity Questionnaire-Short Form. The questionnaire assessing the level of physical activity over the past 7 days provides information about walking, moderate activities, and time spent sitting. Individuals' physical activity levels are divided into three categories according to the scores obtained: "inactive", "minimally active" and "very active".
St. George's Respiratory Questionnaire, SGRQ | baseline to 6 week after
  The quality of life of individuals, a test that measures health-related quality of life for respiratory diseases, ST. George Respiratory Questionnaire. st. George Respiratory Questionnaire; It has three sub-branches as symptoms (8 items), activities (16 items), and effects of the disease (26 items) and consists of a total of 50 items. The total score of the test is between 0-100 (0 score is normal, 100 indicates maximum disability.)
Fatigue Severity Scale | baseline to 6 week after
  The Fatigue Severity Scale, which measures the severity of fatigue in the last month, was used to determine the severity of fatigue. The scale consists of nine questions and each question is graded over seven points. The total score ranges from 9 to 63 points. High scores indicate fatigue, 28 points and above indicate the presence of severe fatigue.
Nottingham Health Profile | baseline to 6 week after
  The Nottingham Health Profile was also used to assess the participants' health-related quality of life. NSP is a general quality of life questionnaire that measures the individual's perceived health problems and the level of these problems that affect normal daily activities. The first part of the NSP, which was developed in two parts, consists of 38 items and evaluates six parameters related to health level.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Nur Demircan, PT, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sun J, He WT, Wang L, Lai A, Ji X, Zhai X, Li G, Suchard MA, Tian J, Zhou J, Veit M, Su S. COVID-19: Epidemiology, Evolution, and Cross-Disciplinary Perspectives. Trends Mol Med. 2020 May;26(5):483-495. doi: 10.1016/j.molmed.2020.02.008. Epub 2020 Mar 21. PMID 32359479
- [Background] MS AG, N.; Surendran, P.; Jacob, P.; Karpouzis, V.; Haneef, M.; Aleef, M.; Ali, S.; Praveen, R.; Bouguerra, E.; Almudahka,. Acute Care Physiotherapy Management of COVID-19 Patients in Qatar: Best Practice Recommendations. Preprints. 2020.
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Gattinoni L, Coppola S, Cressoni M, Busana M, Rossi S, Chiumello D. COVID-19 Does Not Lead to a "Typical" Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2020 May 15;201(10):1299-1300. doi: 10.1164/rccm.202003-0817LE. No abstract available. PMID 32228035